CLINICAL TRIAL: NCT05012319
Title: A Double-Blinded, Placebo-Controlled Parallel, Phase 3 Clinical Efficacy Study Evaluating Nitric Oxide Nasal Spray (NONS) To Treat and Prevent the Exacerbation of Infection in Individuals With Documented Asymptomatic or Mild COVID-19
Brief Title: Phase 3 Clinical Study Evaluating Nitric Oxide Nasal Spray (NONS) Efficacy To Treat and Prevent the Exacerbation of Infection in Individuals With Documented Asymptomatic or Mild COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salmaniya Medical Complex (Other Government)
Responsible Party: Principal Investigator, jameela al salman, infectious disease consultant, Salmaniya Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVIDTX-CTP-07
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, Phase 3 clinical efficacy study evaluating NONS in healthy adult volunteers as a treatment for high-risk asymptomatic and symptomatic individuals with mild COVID-19 infection.
Who Masked: Participant, Care Provider, Investigator
Masking Description: the list of the members of the resrach team who will be blinided have been identiifed and a full procedure has been identified
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Experimental): Nitric Oxide Nasal Spray "Enovid"
  Interventions: Drug: to be given as a treatment
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: to be given as a treatment

INTERVENTIONS:
Drug: to be given as a treatment — Nitric Oxide Nasal Spray "Enovid"

SUMMARY:
Study Design: This is a double-blind, placebo-controlled, Phase 3 clinical efficacy study evaluating NONS in adult volunteers as a treatment for high-risk asymptomatic and symptomatic individuals with mild COVID-19 infection. thru facility).

DETAILED DESCRIPTION:
Study Design: This is a double-blind, placebo-controlled, Phase 3 clinical efficacy study evaluating NONS in adult volunteers as a treatment for high-risk asymptomatic and symptomatic individuals with mild COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* 18 years and above.
* COVID-19 infection Confirmed with a laboratory SARS-CoV-2 RT-PCR nasal swab or antigen test. COVID-19 test specimen must be collected 48 hours prior to Screenings.
* Mild COVID-19 Infection defined as:

  * No Pneumonia (negative by chest auscultation or Chest X Ray).
  * No Shortness of breath.
  * No Tachypnea (respiratory rate <20 breathes/min)
  * No Hypoxia (Oxygen saturation >93% on RA)
  * Fever <38 degrees.
  * No Chest Pain.
  * No Mental Status Change.
* Asymptomatic participants must be high risk defined as (any of the following):

  * Smokers (at least 5 cigarettes per day)
  * BMI (> 40 kg/m2)
  * History of cardiac or chronic lung disease
  * Clotting predisposing conditions (hemophilia, von Willebrand's disease)
  * Sickle cell disease
  * Immunocompromised such as HIV , cancer , on immunosuppressant medications

Exclusion Criteria:

* Participants diagnosed with another (non-COVID-19) respiratory infection.
* Participants with a current tracheostomy or laryngectomy.
* Participants who are receiving concomitant respiratory therapy such as oxygen, positive airway pressure or ventilatory support. NOTE: Positive airway pressure for obstructive sleep apnea is permitted if the treatment was established with good compliance for at least 3 months before study enrollment.
* Participants with newly diagnosed illnesses that are not deemed stable by the participant's primary care physician), based on Investigator assessment of medical history during Screening.
* Participants who use intranasally dosed drugs, prescriptions or over-the-counter medications such as fluticasone.
* Participants who need hospitalization for reasons other than COVID-19 infection.
* Participants who are unable to safely self-administer the nasal spray as directed.
* Clinical signs indicative of moderate, severe, or critical COVID severity symptoms (requirement for supplemental oxygen, limitation of activities due to COVID-19 symptoms).
* Females who are breastfeeding, pregnant, or attempting to become pregnant.
* Participants who have experienced symptoms of COVID-19 for more than 7 days prior to randomization.
* Participants who have any other condition that, in the opinion of the Investigator, would interfere with a participant's ability to adhere to the protocol (eg, participants who are mentally or neurologically disabled and who are considered not fit for their participation in the study), interfere with assessment of the investigational product, or compromise the safety of the participant, or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
efficacy of NONS compared to placebo in participants with COVID-19 to reduce the need of urgent care | 6 months
  To evaluate the efficacy of NONS compared to placebo to reduce the need for urgent medical care in term of the need of visiting the emergency room in participants with COVID-19 infection and reduce of symptoms.

SECONDARY OUTCOMES:
efficacy of NONS compared to placebo in participants with COVID-19 to reduce mortality | 6 months
  To evaluate the efficacy of NONS compared to placebo to reduce mortality of participants with COVID-19
efficacy of NONS compared to placebo in participants with COVID-19 on viral load reduction | 6 months
  Viral load reduction measure in copies per ml in participants with mild COVID-19 infection.
efficacy of NONS compared to placebo in participants with COVID-19 to reduce time of clinical symptoms improvement | 6 months
  Median time reduction to COVID-19 clinical symptoms improvement in days
Incidence of Treatment-Emergent Adverse Events | 6 months
  Incidence of Treatment-Emergent Adverse Events to assess Safety and Tolerability]

CONTACTS AND LOCATIONS:
Locations (1):
- Abdulla Kanoo Center,, A'ali, Building 556, Bahrain